CLINICAL TRIAL: NCT00248729
Title: Etomidate Versus Midazolam for Pre-Hospital Intubation: A Prospective, Randomized Trial
Brief Title: Effectiveness and Safety Study of Etomidate Versus Midazolam to Help Place a Breathing Tube Outside of the Hospital.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Luke's Hospital, Pennsylvania (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: SLHN 001
Record Dates: First submitted 2005-11-02; First posted 2005-11-04 (Estimated); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Etomidate; Midazolam

INTERVENTIONS:
Drug: Etomidate (20mg) or Midazolam (7mg)

SUMMARY:
The objective of this study was to compare the utility of etomidate and midazolam in helping patients to relax when there was a need for the placement of a ventilation tube by medics who were transporting patients to a hospital in an ambulance.

DETAILED DESCRIPTION:
Study Objective: The objective of this study was to compare the utility of etomidate and midazolam for sedative facilitated intubation (SFI), without paralytics, in pre-hospital adult patients.

Methods: This prospective, double-blind, randomized trial was conducted with two ground pre-hospital Advanced Life Support (ALS) units. All patients age 18 or over transported by the two participating systems requiring pre-hospital SFI were eligible for participation. The ambulances were stocked with blinded numbered syringes, each containing either 7mg of midazolam or 20mg of etomidate. Contact with the Medic Command physician was not required and no paralytics were used. If sedation was not achieved with the study drug, medics could request additional sedation from a Medical command physician; only midazolam or diazepam were available outside of the study.

ELIGIBILITY:
Inclusion Criteria:

Under the study protocol, all patients age 18 or over transported by the two participating ALS systems, requiring pre-hospital Sedation Facilitated Intubation, were eligible for participation.

Exclusion Criteria:

Exclusion criteria were pregnancy and age less than 18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-10; Study Completion 2005-11

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne L Jacoby, MD, Principal Investigator — St. Luke's Hospital
Locations (1):
- St. Luke's Hospital, Bethlehem, Pennsylvania, United States